CLINICAL TRIAL: NCT06215482
Title: The Effect of "Adjacent Bed Effect" Induced by Anxiety on the Perioperative Period of Patients With Chocolate Cyst of Ovary
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2024-07-201
Record Dates: First submitted 2024-01-07; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Participants' Pain,Quality of Life and Hospital Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- "A-N" group (Anxious-Non-anxious group): Upon admission, participants filled out a Anxiety Disorder Screening Scale, this group scored <10 points
- "N-N" group (Non-anxious-Non-anxious group): Upon admission, participants filled out a Anxiety Disorder Screening Scale, this group scored ≥10 points

SUMMARY:
The "adjacent bed effect" caused by anxiety leads to poor recovery of participants after ovarian chocolate cyst surgery, including pain and quality of life, and affects participant satisfaction with the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Ovarian chocolate cyst diameter ≥4cm;
2. Infertility;
3. Dysmenorrhea medications were ineffective; Any one of the above, with or without clinical symptoms.

Exclusion Criteria:

1. Age <18 years old;
2. Previous history of other surgeries;
3. Previous history of nervous system diseases, such as Parkinson's disease, dementia, etc.
4. Previous history of blood system diseases, such as leukemia;
5. Unable to tolerate surgery due to serious complications, such as serious cardiovascular and cerebrovascular diseases;
6. Inability to complete the questionnaire due to language or learning disabilities;
7. Those who don't want to participate.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anxious or nonanxious state in participants with chocolate cysts
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-07-22 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-23 (Actual)

PRIMARY OUTCOMES:
participant demographic information | through study completion, an average of 2 month
  A self-rating anxiety scale was filled out and part of the participant's clinical information was collected,higher scores indicate more anxiety; Maximum 100 and minimum 0

SECONDARY OUTCOMES:
Postoperative Scale scores | through study completion, an average of 2 month
  visual analogue scale were completed after operation; higher scores indicate more pain;Maximum 100 and minimum 0
scale were completed after operation | through study completion, an average of 2 month
  Numerical Rating Scale for Pain scale were completed after operation;higher scores indicate more pain;Maximum 100 and minimum 0
scale were completed after operation | through study completion, an average of 2 month
  Quality of Life Scale for patients with endometriosis were completed after operation; higher scores indicate worse quality of life;Maximum 100 and minimum 0
scale were completed after operation | through study completion, an average of 2 month
  hospital satisfaction scale were completed after operation higher scores indicate more satisfied with the hospital; Maximum 100 and minimum 0

CONTACTS AND LOCATIONS:
Overall Officials: Qiong joan_zhang2002@sina.com, Study Chair — Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University
Locations (1):
- Qiong Zhang, Wenzhou, China